CLINICAL TRIAL: NCT02189616
Title: Evaluate the Clinical Efficacy of Mobile Phone Short Message Service (SMS) Reminder and Consultation on the Self-management and Outcomes of Poorly-controlled Asthma: a Multicenter Randomized Controlled Trial
Brief Title: Efficacy of Mobile Phone Short Message Service (SMS) Reminder and Consultation on Asthma Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Baoji Central Hospital (Other); Hanzhong Central Hospital (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Principal Investigator, songlq, vice director of department of respirotary and critical care medine, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xjhx-song2
Record Dates: First submitted 2014-03-24; First posted 2014-07-14 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
Keywords: asthma management; SMS reminder; SMS consultation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- regular care group (Other): receive regular care which contains filling a paper asthma diary daily.
  Interventions: Other: regular care
- SMS reminder group (Experimental): receive weekly mobile phone short message reminders for 3 months
  Interventions: Behavioral: SMS reminder; Other: regular care
- SMS reminder and SMS consultation group (Experimental): receive weekly mobile phone short message reminders and can consult asthma nurse by mobile phone short message when needed for 3 months
  Interventions: Behavioral: SMS reminder; Other: SMS consultation; Other: regular care

INTERVENTIONS:
Behavioral: SMS reminder — send weekly mobile phone short message reminders to the intervention group
  Arms: SMS reminder and SMS consultation group; SMS reminder group
Other: SMS consultation — told patients to consult qualified asthma nurses by SMS when they need
  Arms: SMS reminder and SMS consultation group
Other: regular care — patients are asked to fill in their paper asthma diary daily for 3 months

SUMMARY:
Asthma is the disease being studied. The main objective of this study is to assess the clinical efficacy of mobile phone short message service (SMS) reminder and consultation on the self-management and outcomes of poorly controlled asthma which is first diagnosed in a time period of 3 months. The secondary objective is to explore the cost-benefit and cost-effectiveness of the proposed intervention.

Aims: The main aim of this study is to assist asthma patients to practice asthma self-management at home by sending reminders and responding to patients' consultations with mobile phone short message service (SMS), which will eventually help them to control their asthma, and prevent asthma exacerbation. Thus, the ultimate goal of this proposed study is to improve patient health outcome via enhancing patient-physician interaction through mobile phone short message service (SMS) that is low-cost and could be followed easily by the patients and their physicians.

The hypothesis is that asthma patients who receive weekly text message reminders to educate them and reinforce adherence will have better asthma outcome, such as asthma control, while the intervention integrating patient consultation and reminders by SMS improve asthma outcome even more. The investigators further hypothesize that these subjects under intervention will have an improvement in secondary measures including quality of life and patient satisfaction. The investigators also anticipate that such an approach in asthma management will be cost-effective.

DETAILED DESCRIPTION:
After examined for their eligibility and recruited into this study at outpatient service, all participants have their case records which contain their baseline data and receive the same standard asthma education(including basic knowledge about asthma, how to use their medicine, what to do when an asthma attack happens and when to come back for their disease review and so on). Each patient is given a paper asthma diary and a peak expiratory flow(PEF) measurer for free. In addition, they are told what intervention they will receive and revised face-to-face one month after the beginning of intervention. After the 3-month study period, when they return to the hospitals, they will return the asthma diaries, be asked to fill in the questionnaires and take pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosed uncontrolled or partly-controlled asthma by Global Initiative for Asthma(GINA) standard.
2. At least 6 months asthma history.
3. Ownership of a mobile phone and currently using the text messaging service.
4. Age between 18 and 65 years old.
5. Willingness to participate in this study.
6. Willing to sign the written informed consent to take part in the study.

Exclusion Criteria:

1. Inability to provide written informed consent or to fill in the paper asthma diary.
2. A history of smoking cigarettes for greater than ten pack years.
3. Other current or a history of severe comorbidity.
4. Being in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
change in asthma control measured by Asthma Control Test(ACT) | 3 months
  change in asthma control measured by Asthma Control Test(ACT) between baseline and 3 months after randomization.
score of knowledge, attitude, and self efficacy asthma questionnaire (KASE-AQ) | 3 months
  score of knowledge, attitude, and self efficacy asthma questionnaire (KASE-AQ) at baseline and 3 months

SECONDARY OUTCOMES:
Mini-asthma quality of life questionnaire (mini-AQLQ) | 3 months
  mini-AQLQ scores at baseline and 3 months after the randomization
asthma control | 3 months
  change of asthma control level indicated by symptom score, PEF and asthma exacerbations (asthma hospitalizations, emergency department visits, or oral corticosteroid dispensing) from baseline to the end of intervention(3 months)

OTHER OUTCOMES:
cost effectiveness | 3 months
  The cost effectiveness of SMS reminder and consultation interventions compared to controls without study interventions.

CONTACTS AND LOCATIONS:
Overall Officials: liqiang song, doctor, Principal Investigator — first affiliated hospital, the fourth military medical university
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China